CLINICAL TRIAL: NCT02316184
Title: Comparing Brief Alcohol Interventions For HIV-HCV Co-infected Persons
Acronym: REACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Responsible Party: Principal Investigator, Michael Stein, MD, Principal Investigator (MPI), Butler Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AA023726
Record Dates: First submitted 2014-12-10; First posted 2014-12-12 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: HIV; Hepatitis C
Keywords: Alcohol
MeSH Terms: conditions — Hepatitis C | interventions — Motivational Interviewing; Crisis Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brief Advice (Placebo Comparator): Participants in this arm will receive brief advice about alcohol use. Sessions will occur at the baseline interview and every three months for 18 months.
  Interventions: Behavioral: Brief Advice
- MI (Active Comparator): Participants in this arm will receive a talking intervention designed to explore their interest in reducing/eliminating alcohol use. Sessions will occur at the baseline interview and every three months for 18 months.
  Interventions: Behavioral: Motivational Interviewing

INTERVENTIONS:
Behavioral: Motivational Interviewing — Motivational Interviewing is a client-centered method of exploring individual's interest in making behavioral changes. In this study, the targeted behavior is alcohol use.
  Arms: MI
Behavioral: Brief Advice
  Arms: Brief Advice

SUMMARY:
Two types of brief intervention, Brief Advice (BA) and Motivational Interviewing (MI), have been shown to be efficacious in reducing drinking in non-HIV samples. Our goal is to determine whether offering counseling beyond Brief Advice, namely MI, has greater alcohol reduction effects. In the proposed randomized trial, all 300 HIV-HCV co-infected participants will receive BA delivered by their HIV PCP during a regular HIV visit and will then be randomized to either a 30-minute Motivational Interviewing Intervention with a Behavioral Counselor (MI) or to HIV clinic treatment-as-usual. After this initial meeting, drinking "check-in" (MI or BA) sessions will then be provided telephonically every three months for 18 months, with a final assessment at 24 months. Our primary outcome is drinks per week.

DETAILED DESCRIPTION:
Two types of brief intervention, Brief Advice (BA) and Motivational Interviewing (MI), have been shown to be efficacious in reducing drinking in non-HIV samples. Our goal is to determine whether offering counseling beyond Brief Advice, namely MI, has greater alcohol reduction effects. In the proposed randomized trial, all 300 HIV-HCV co-infected participants will receive BA delivered by their HIV PCP during a regular HIV visit and will then be randomized to either a 30-minute Motivational Interviewing Intervention with a Behavioral Counselor (MI) or to HIV clinic treatment-as-usual. After this initial meeting, drinking "check-in" (MI or BA) sessions will then be provided telephonically every three months for 18 months. Research assessments will also be done every three months, with a final assessment at 24 months. Our primary outcome is drinks per week.

ELIGIBILITY:
Inclusion Criteria:

* HIV+
* HCV RNA positive
* consuming on average at least 4 alcoholic drinks per week in the last month
* 18 years or older

Exclusion Criteria:

* current, severe psychiatric symptoms requiring immediate clinical attention (e.g., suicidal ideation, current mania, psychosis)
* inability to understand English
* cognitive impairment severe enough to interfere with ability to actively participate
* hepatocellular carcinoma or life expectancy less than 24 months
* plan to move from Providence area in the next 24 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
Alcohol Use questionnaire | up to 24 months
  participants will be asked how many drinks/week they have

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stein, MD, Principal Investigator — Butler Hospital
Locations (2):
- United States (2):
  - Butler Hospital, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island

REFERENCES:
- [Derived] Stein MD, Herman DS, Kim HN, Howell A, Lambert A, Madden S, Moitra E, Blevins CE, Anderson BJ, Taylor LE, Pinkston MM. A Randomized Trial Comparing Brief Advice and Motivational Interviewing for Persons with HIV-HCV Co-infection Who Drink Alcohol. AIDS Behav. 2021 Apr;25(4):1013-1025. doi: 10.1007/s10461-020-03062-2. Epub 2020 Oct 12. PMID 33047258